CLINICAL TRIAL: NCT05702619
Title: Hypoxia-driven Prostate Cancer Genomics (HYPROGEN) - Illuminating the Genomic Landscape of Hypoxia-driven Early Metastatic Prostate Cancer
Brief Title: Hypoxia-driven Prostate Cancer Genomics (HYPROGEN)
Acronym: HYPROGEN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Prostate Cancer UK (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp155
Record Dates: First submitted 2022-11-03; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer; Hypoxia
Keywords: genomic; multi-omic
MeSH Terms: conditions — Prostatic Neoplasms; Hypoxia | interventions — Circulating Tumor DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of bone samples and prostate biopsy samples and multi-omic analysis including genomics
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1: Arm 1 - De novo, treatment-naïve metastatic prostate cancer
  Interventions: Drug: Optional non-IMP pimonidazole; Diagnostic Test: CT-guided Bone Biopsy; Diagnostic Test: TRUS-guided Targeted Transperineal Prostate Biopsy; Diagnostic Test: Whole-body MRI; Other: Baseline bloods - for germline testing; Other: Baseline bloods for CTCs and ct DNA taken at same time as baseline bloods in Arm 1; Other: Post-pimonidazole bloods for CTCs and ctDNA
- Arm 2: Arm 2 - De novo, treatment- naïve localised prostate cancer planned for radical prostatectomy
  Interventions: Drug: Optional non-IMP pimonidazole; Procedure: Radical Prostatectomy; Diagnostic Test: Prostate MRI scans; Other: Baseline bloods - for germline testing

INTERVENTIONS:
Drug: Optional non-IMP pimonidazole — patients will be asked to ingest an oral formulation of pimonidazole hydrochloride (HCl) (Oral HypoxyprobeTM-1). Pimonidazole HCl is a marker for hypoxia in tumour tissue when ingested as an encapsulated solid. Following oral administration, pimonidazole distributes throughout the body where it covalently binds to normal and tumour tissues that have regions of low oxygen concentrations (pO2 of ≤ 10 mmHg at 37oC). The tissue binding can be visualised by immunohistochemistry / light microscopy. The capsules are to be taken within 8-16 hours (optimal timepoint 12 hours) before the planned first biopsy within Arm 1 and before radical prostatectomy for patients in Arm 2. If the patient refuses the pimonidazole, forgets to take it, or if it is not available, the patient can still participate in the study and their samples will be stained for hypoxia post-biopsy.
  Other Names: Pimonidazole Hydrochloride
Diagnostic Test: CT-guided Bone Biopsy — A CT-guided biopsy of a bone metastasis that is deemed to be easy to biopsy and in an area without major risk for pathological fracture or bleeding will be taken during the biopsy visit. Patients will receive routine local anaesthetic of the region to be biopsied followed by thorough disinfection of the biopsy site with antiseptic wipes. Patients will be asked to fast on the day of the procedure and to have an intravenous cannula inserted to allow the use of medication causing minimal sedation (for example midazolam and/or fentanyl) during the procedure if required to alleviate discomfort or pain.
  Groups: Arm 1
Diagnostic Test: TRUS-guided Targeted Transperineal Prostate Biopsy — Transperineal Prostate Biopsy will be performed following standard clinical practice of local department. This will include pre-operative oral analgesia and prophylactic antibiotic treatment according to local hospital policy for transperineal prostate biopsies.
  Groups: Arm 1
Procedure: Radical Prostatectomy — Radical Prostatectomy will be performed according to standard of care robotic approach and as relayed to the patient by the attending urologic surgeon. The side effects of the surgery are the ones reported in the literature and the latest participant information leaflet provided prior patient consent (e.g. risk of erection disfunction, incontinence, etc.).
  Groups: Arm 2
Diagnostic Test: Whole-body MRI — Whole-body MR imaging (wbMRI) will be performed once, before or after the biopsy study visit, depending on available examination slots in the Department of Radiology. WbMRI images will allow comparison of the numbers of bone metastases detected by routine bone scan and wbMRI for sensitivity assessment of both techniques for oligometastatic disease.
  Groups: Arm 1
Diagnostic Test: Prostate MRI scans — Patients within Arm 2 will be offered the option to undergo additional MR imaging of the pelvis in addition to any standard of care imaging acquired. In patients who agree to undergo additional scans, MRI scans will be performed on 2 occasions prior to the radical prostatectomy. MRI scans will be acquired on either the MR sim diagnostic scanner, on the MR Linac scanner or on both.
  Groups: Arm 2
Other: Baseline bloods - for germline testing — Arm 1 -
  * 1-2 x 3.5mL blood samples collected into EDTA tubes for germ line DNA extraction and processing to PBMC for banking and future profiling of immune cell populations
  * 1 x 10mL serum tubes for future, biobank related research projects, ie lipidomics, metabolics and microRNA analysis
  ARM 2 -
  A blood sample (maximum 20ml) will be taken for standard of care blood tests prior to prostatectomy including Full Blood Count, Renal Function and PSA. At the same time these standard of care bloods are taken, additional bloods - a maximum of 30ml - will be taken for research purposes as required for the following downstream analysis:
  * Germ line DNA extraction and optional processing to PBMC for banking and future profiling of immune cell populations
  * Biobank related research projects, ie lipidomics, metabolics and microRNA analysis
Other: Baseline bloods for CTCs and ct DNA taken at same time as baseline bloods in Arm 1 — 2 x 10mL Streck cell-free DNA blood collection tubes® for circulating tumour cell (CTC) collection and circulating tumour DNA (ctDNA) extraction.
  Groups: Arm 1
Other: Post-pimonidazole bloods for CTCs and ctDNA — ARM 1 - 2 x 10mL Streck cell-free DNA blood collection tubes® for circulating tumour cell (CTC) collection and circulating tumour DNA (ctDNA) extraction.
  Groups: Arm 1

SUMMARY:
Due to the rapid growth, tumour demand for oxygen is often higher than what can be delivered by the newly forming blood vessels. Tumour adaption to this imbalanced oxygen supply and demand (hypoxia) is associated with poor prognosis and genetic changes (genomic instability) that allow it to become more resistant to chemo- and radiotherapy. Patients with hypoxic tumours therefore die earlier. Limited information is available on hypoxia in newly diagnosed prostate cancer, especially to what degree hypoxia in the prostate tumour is associated with the presence of metastases to bones. The Hyprogen trial is a prospective, non-randomised, exploratory biopsy and imaging biomarker study recruiting 60 patients with prostate cancer to better establish the role of hypoxia in prostate cancer cells evolution and early metastatic spread.

DETAILED DESCRIPTION:
Arm 1 of this study will aim to determine the association between hypoxia in the primary tumour with the presence of skeletal metastases and aim to determine if hypoxia is also present in the metastatic sites themselves. Arm 2 will aim to determine the genetic changes associated with hypoxia in cancers that have not spread outside the prostate. Hypoxia presence will be determined by using a hypoxia identifying stain (by giving a patient a tablet of the stain to take orally) and by identifying genomic alterations that are associated with hypoxia. After taking the tablet of the hypoxia marker (Pimonidazole) patients in Arm 1 will receive both a biopsy of the prostate and of one or two of the bone metastases. The presence or not as well as the degree of hypoxia in both sites will be assessed. Patients in Arm 2 will receive pimonidazole prior to a planned radical prostatectomy and the heterogeneity of hypoxia related genetic change throughout the prostate will assessed. Arm 2 patients will undergo MRI hypoxia imaging to validate the detection of pimonidazole marked hypoxic regions with a non-invasive imaging method.

ELIGIBILITY:
ARM 1

Inclusion Criteria:

* Male patients aged 18 years and older
* Histologically proven adenocarcinoma of the prostate (≥cT2) or Highly suspected metastatic prostate cancer
* PSA value of ≥ 20 ng/mL
* Multiple lesions (≥ 5) suspicious of metastatic spread on routine imaging procedures with at least one amenable* to biopsy (cohort A) or oligometastatic bone disease (≥1 to ≤ 4) at routine bone scan with at least one lesion amenable* to biopsy (cohort B)

  *e.g. safely to biopsy and expectably providing sufficient tissue yield World Health Organisation (WHO) performance status 0 to 2 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 months
* No prior local and/or systemic treatment for localised prostate cancer
* Willing to donate cancer tissue samples for research purposes (bone metastasis and primary tumour)

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to staff at the study site)
* Previous enrolment in the HYPROGEN study
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g. uncompensated respiratory, cardiac, hepatic or renal disease)
* Evidence of any other significant clinical disorder or laboratory finding that made it undesirable for the patient to participate in the study
* Any investigational agents or study drugs from a previous clinical study within 30 days of the first tissue collection
* Prior treatment of localized prostate cancer including radiotherapy and/or androgen-deprivation therapy
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
* Contra-indications to MRI (incl. pacemakers etc.)
* Bone metastases in difficult to reach areas or areas which might be at risk for pathological fracture post biopsy as judged by biopsying radiologist / chief investigator
* Increased risk of bleeding as a result of biopsy
* History of bleeding disorders or thrombocytopenia (platelets <100/nL)
* Concomitant treatment with anticoagulant therapy, e.g. warfarin/low molecular weight heparin or Anti-Xa-inhibitors and other NOACs, if temporary cessation medically not justifiable
* Current urinary tract infection (UTI) or prostatitis

ARM 2

Inclusion Criteria:

* Male patients aged 18 years and older cT¬2-T3 / cN0-N1 / cM0 Any Group Grade (GG) 2-5: this includes Gleason scores 3+4, 4+3, 4+4, 4+5, 5+3, 5+4, 5+5. Any PSA
* Histologically proven adenocarcinoma of the prostate
* Undergoing radical prostatectomy as primary treatment for localised prostate cancer
* World Health Organisation (WHO) performance status 0 to 2 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 months
* No prior local and/or systemic treatment for localised prostate cancer
* Willing to donate cancer tissue samples for research purposes (any metastasis and primary tumour)

Exclusion criteria:

* Involvement in the planning and/or conduct of the study (applies to staff at the study site)
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g. uncompensated respiratory, cardiac, hepatic or renal disease)
* Any investigational agents or study drugs from a previous clinical study within 30 days of the first tissue collection
* Prior treatment of localized prostate cancer including radiotherapy and/or androgen-deprivation therapy
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
* Contra-indications to MRI (incl. pacemakers etc.)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Arm 1 - De novo, treatment-naïve metastatic prostate cancer Arm 2 - De novo, treatment- naïve localised prostate cancer planned for radical prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-10-03 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure | 24 months
  To document the differential genomic aberrations and gene expressional alterations in hormone-naïve primary prostate cancers and paired skeletal metastases with respect to the presence or abscence of tissue hypoxia in the tumour samples.

SECONDARY OUTCOMES:
Secondary outcome measure | 24 months
  To determine extent of CTCs DNA in treatment naive metastatic prostate cancer in the presence or absence of hypoxia

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

DOCUMENTS (1):
  • Study Protocol (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT05702619/Prot_000.pdf